CLINICAL TRIAL: NCT05125861
Title: Dynamic Cerebral Autoregulation of Remote Ischemic Conditioning Combined With Intravenous Thrombolysis for Acute Ischemic Stroke
Acronym: CARIC-IVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARIC-IVT
Record Dates: First submitted 2021-11-01; First posted 2021-11-18 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Remote Ischemic Conditioning
Keywords: Remote Ischemic Conditioning; Dynamic Cerebral Autoregulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Active Comparator): RIC+Standard medical treatment Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mmHg. RIC will be conducted twice within 6 to 24 hours from thrombolysis.
  Interventions: Procedure: remote ischemic conditioning
- control group (Placebo Comparator): Sham RIC+Standard medical treatment Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mmHg. RIC will be conducted twice twice within 6 to 24 hours from thrombolysis.
  Interventions: Procedure: sham remote ischemic conditioning

INTERVENTIONS:
Procedure: remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mmHg. All patients underwent dynamic cerebral autoregulation on days 1-2 and 7-10 after onset, and intravenous blood was collected by a nurse and stored in the laboratory 0-6 hours after thrombolysis and 24 hours after thrombolysis.
  Arms: RIC group
Procedure: sham remote ischemic conditioning — Sham remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mmHg. All patients underwent dynamic cerebral autoregulation on days 1-2 and 7-10 after onset, and intravenous blood was collected by a nurse and stored in the laboratory 0-6 hours after thrombolysis and 24 hours after thrombolysis.
  Arms: control group

SUMMARY:
The purpose of this study is to determine the impact of remote ischemic conditioning on dynamic cerebral autoregulation in patients with acute ischemic stroke receiving intravenous thrombolysis.

DETAILED DESCRIPTION:
In this study, cases of ischemic stroke who undergo intravenous thrombolysis within 4.5 hours from onset are included. The experimental group receive basic treatment and remote ischemic conditioning for 200mmHg, 2 times within 6 hours to 24 hours from thrombolysis. The control group receive basic treatment and remote ischemic conditioning control for 60mmHg, 2 times within 6 hours to 24 hours from thrombolysis . Both groups underwent dynamic cerebral autoregulation measurements at days 1 to 2 and 7 to 10 of onset and recorded the relevant indexes, and blood samples were collected before and 24 hours after intravenous thrombolysis, we aimed to determine the impact of remote ischemic conditioning combined with intravenous thrombolysis on dynamic cerebral autoregulation in acute ischemic stroke patients. We hypothesized that remote ischemic conditioning would improve dynamic cerebral autoregulation in patients with acute ischemic stroke receiving intravenous thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years, < 80 years, regardless of sex;
2. Patients with clinically definite diagnosis of acute ischemic stroke and undergo intravenous thrombolysis;
3. Baseline NIHSS >= 5, and <= 25;
4. Baseline GCS ≥8;
5. Signed and dated informed consent is obtained

Exclusion Criteria:

1. Patients who undergo endovascular treatment;
2. mRS ≥ 2 before the onset of the disease;
3. Severe organ dysfunction or failure;
4. Those who have a history of atrial fibrillation;
5. The patients who have the contraindication of remote ischemic conditioning treatment, such as severe soft tissue injury, fracture or vascular injury in the upper limb, acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc;
6. Pregnant or lactating women;
7. Patients with a life expectancy of less than 3 months or patients unable to complete the study for other reasons;
8. He/She is participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to admission;
9. Other conditions that the researchers think are not suitable for the group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Dynamic cerebral autoregulation of affected sides measured by phase difference(PD) in Degree | 1-2 days
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.

SECONDARY OUTCOMES:
Dynamic cerebral autoregulation of unaffected sides measured by phase difference(PD) in Degree | 1-2 days
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.
Dynamic cerebral autoregulation of affected sides measured by phase difference(PD) in Degree | 7-10 days
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.
Dynamic cerebral autoregulation of unaffected sides measured by phase difference(PD) in Degree | 7-10 days
  A dynamic cerebral auto-regulation parameter derived from transfer function analysis.Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.
Hematology related indicators | before and 24 hours after intravenous thrombolysis
  Blood samples were collected before and 24 hours after intravenous thrombolysis

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China